CLINICAL TRIAL: NCT04962854
Title: Changes of Bone Mineral Density in Total Hip Arthroplasty - A Prospective Comparison of Isoelastic and Metal-backed Cup Designs
Brief Title: Changes of Bone Mineral Density in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: St. Vincent Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Michael Tiefenboeck, Dr. med. univ, St. Vincent Hospital, Vienna
Other Study IDs: DEXA THA
Record Dates: First submitted 2021-07-10; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Bone Mineral Density
Keywords: Total Hip Arthroplasty; DEXA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Monoblock Cup: 53 patients received a monoblock cup (RM Pressfit vitamys®)
- Modular Cup: 64 patients received a modular cup (ANA.NOVA® Implantec)

SUMMARY:
The study was performed as a prospective, single center study at the Department of Orthopedics, Sacred Heart of Jesus Hospital Vienna, Austria. 117 patients were enrolled in a from January 2016 to May 2017. 53 patients received an isoelastic monoblock cup (RM Pressfit vitamys® Mathys) and 64 patients received a metal- backed modular cup (ANA.NOVA® ImplanTec). Dual-energy x-ray absorptiometry scans according to DeLee and Charnley Zones were performed at time points 0, 3, 6, 12, and 24 months after surgery. The aim of thise study was to compare changes in BMD between an isoelastic monoblock cup and a titanium modular cup. We hypothesized that the more elastic monoblock cup performs better than the more rigid modular cup with regard to changes in BMD.

DETAILED DESCRIPTION:
The study was performed as a prospective, single center study at the Department of Orthopedics, Sacred Heart of Jesus Hospital Vienna, Austria.

Inclusion criteria were as follows: any patient aged from 18 years onwards undergoing primary cementless THA for degenerative joint disease, including osteoarthritis, post-traumatic arthritis, congenital hip dysplasia and avascular necrosis. Excluded were all patients with malignant diseases and pregnant women, additionally, patients were excluded if severe complications such as fracture or revision surgery occurred during the study period.

Patients were enrolled from January 2016 to May 2017, a total of 117 patients were included. All patients underwent uncemented THA, patients either received a monoblock cup (RM Pressfit vitamys®; Mathys Ltd. Bettlach, Switzerland), or a titanium shell (ANA.NOVA® Implantec, Mödling, Austria). DEXA measurements according to the DeLee and Charnley Zones were performed postoperatively, 3, 6, 12 and 24 months after primary hip arthroplasty. Bone mineral density (BMD) was measured by using the bone densiometer (Lunar, Prodigy, GE Medical Sytsems). A special legholder was used to fix the leg to ensure the same rotation and avoid measurement errors. DEXA measurements were performed and analyzed by two trained authors. Statistical analysis focused on differences in BMD between monoblock cup and modular cup after 3, 6, 12 and 24 months as well as changes in BMD in relation to cup inclination. In order to gain valid results, the nonparametric Wilcoxon rank-sum test was used. We used t-Test to evaluate differences to the baseline. A probability value of p ≤0.05 was considered as statistically significant. Data was analyzed using Microsoft Excel® and SPSS® (version 26.0, SPSS Inc., Chicago, IL, USA) representing standard statistical software. We hypothesized that the more elastic monoblock cup performs better than the more rigid modular cup with regard to changes in BMD.

ELIGIBILITY:
Inclusion Criteria:

* any patient aged from 18 years onwards undergoing primary cementless THA for degenerative joint disease, including osteoarthritis, post-traumatic arthritis, congenital hip dysplasia and avascular necrosis.

Exclusion Criteria:

* patients with malignant diseases and pregnant women, additionally, patients were excluded if severe complications such as fracture or revision surgery occurred during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who either received a monoblock cup (RM Pressfit vitamys®; Mathys Ltd. Bettlach, Switzerland), or a titanium shell (ANA.NOVA® Implantec, Mödling, Austria) between January 2016 and May 2017. 117 patients (female 69, male 48), mean age was 68 years (range, 43 to 89 years)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Dexa meassurments | 24 Months
  Changes in BMD according to DeLee and Charnley Zones

IPD SHARING:
Plan to Share IPD: No